CLINICAL TRIAL: NCT01266343
Title: Comparison of Anterior Chamber Paracentesis and Conventional Mannitol Infusion in Patients With Primary Acute Angle-closure Glaucoma
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Hui-Chun Ho, Department of Ophthalmology, Wanfang Hospital
Other Study IDs: 99018
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Glaucoma; Acute Primary Angle-closure Glaucoma
Keywords: Glaucoma; anterior chamber paracentesis; conventional Mannitol infusion
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental Group
- Control Group

SUMMARY:
The investigators wanted to reported the results of immediate anterior chamber paracentesis (ACP), compared to Mannitol infusion, in patients with acute primary angle-closure glaucoma (PACG). In this study, the investigators first divided patients into three sub-groups according to their initial intraocular pressure (IOP) for analyzing the differences of IOP control, severity of corneal edema, waiting time for laser peripheral iridotomy (LPI), and visual outcome between ACP and Mannitol infusion.

DETAILED DESCRIPTION:
The investigators demonstrated that ACP could be first considered in patients with initial IOP between 45 to 60 mmHg because it provided better visual outcome than Mannitol infusion through the rapid stabilization of the anterior segment, which was achieved by rapid IOP control, better corneal edema regression, shortening waiting time for LPI. However, ACP should be considered in patients with the initial IOP of 60mmHg and higher only when Mannitol was contraindicated.

ELIGIBILITY:
Inclusion Criteria:

* first attack of acute PACG;
* initial presenting IOP was higher than 45 mmHg;
* diagnosis confirmed by gonioscopic examination;
* patients within 48 hours of symptom onset.

Exclusion Criteria:

* been incompletely followed up within 2 weeks;
* been using anti-glaucomatous medication before ACP or Mannitol infusion;
* previous intraocular surgeries on the same eye;
* contraindication for Mannitol;
* history of other vision-threatening ocular diseases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-01; Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chun Ho, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan